CLINICAL TRIAL: NCT06016738
Title: A Phase 3 Randomized, Open-Label Study of OP-1250 Monotherapy vs Standard of Care for the Treatment of ER+, HER2- Advanced or Metastatic Breast Cancer Following Endocrine and CDK 4/6 Inhibitor Therapy (OPERA-01)
Brief Title: OP-1250 (Palazestrant) vs. Standard of Care for the Treatment of ER+/HER2- Advanced Breast Cancer
Acronym: OPERA-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-1250-301; OPERA-01 (Other: Olema Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-08-17; First posted 2023-08-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; ER Positive Breast Cancer; HER2 Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palazestrant (OP-1250) (Experimental): Participants will receive Palazestrant
  Interventions: Drug: Palazestrant
- Standard of Care Endocrine Therapy (Active Comparator): Participants will receive Investigator's choice of one of the Standard of Care drugs (fulvestrant, anastrozole, letrozole, or exemestane)
  Interventions: Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane

INTERVENTIONS:
Drug: Palazestrant — Participants will be treated with palazestrant once daily on a 4 week (28 day) cycle. Doses evaluated in the dose-selection part will be 120 mg once daily and 90 mg once daily.
  Other Names: OP-1250
  Arms: Palazestrant (OP-1250)
Drug: Fulvestrant — Participants will be treated with fulvestrant on C1D1, C1D15, and then on Day 1 of every subsequent 4 week (28 day) cycle
  Arms: Standard of Care Endocrine Therapy
Drug: Anastrozole — Participants will be treated with anastrozole once daily on a 4 week (28 day) cycle
  Arms: Standard of Care Endocrine Therapy
Drug: Letrozole — Participants will be treated with letrozole once daily on a 4 week (28 day) cycle
  Arms: Standard of Care Endocrine Therapy
Drug: Exemestane — Participants will be treated with exemestane once daily on a 4 week (28 day) cycle
  Arms: Standard of Care Endocrine Therapy

SUMMARY:
This phase 3 clinical trial compares the safety and efficacy of palazestrant (OP-1250) to the standard-of-care options of fulvestrant or an aromatase inhibitor in women and men with breast cancer whose disease has advanced on one endocrine therapy in combination with a CDK4/6 inhibitor.

DETAILED DESCRIPTION:
This is an international, multicenter, randomized, open-label, active-controlled, phase 3 clinical trial. The purpose of this trial is to compare the safety and efficacy of palazestrant (OP-1250) as a single agent to the standard of care endocrine therapy: either fulvestrant or an aromatase inhibitor (anastrozole, letrozole, or exemestane).

This trial is seeking adult participants with ER+, HER2- advanced or metastatic breast cancer whose disease has relapsed or progressed on 1 or 2 prior lines of standard-of-care endocrine therapy for metastatic breast cancer. Prior lines of therapy must include one line of endocrine therapy in combination with a CDK 4/6 inhibitor. In the dose-selection part of the trial, approximately 120 participants will be randomized to one of the two doses of palazestrant or to the standard-of-care endocrine therapy. Thereafter, approximately 390 participants will be randomized to palazestrant at the selected dose or to the standard-of-care endocrine therapy.

ELIGIBILITY:
Key inclusion criteria:

* Adult female or male participants.
* ER+, HER2- locally advanced or metastatic breast cancer that is not amenable to curative therapy.
* Evaluable disease (measurable disease or bone-only disease).
* Previously received a CDK4/6 inhibitor in combination with an endocrine therapy in the advanced setting. One additional line of ET as a monotherapy is allowed. Duration of the most recent prior ET must be at least 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic, and renal functions.
* Female participants can be pre-, peri- or postmenopausal.
* Male and pre- or peri-menopausal female participants must be willing to take a GnRH (or LHRH) agonist.

Key exclusion criteria:

* Symptomatic visceral disease, imminent organ failure, or any other reason that makes the participant ineligible for endocrine monotherapy.
* Previously received chemotherapy in the advanced/metastatic setting.
* Previously received treatment with elacestrant or an investigational estrogen receptor-directed therapy.
* History of allergic reactions to study treatment.
* Any contraindications to the selected standard-of-care endocrine therapy in the local prescribing information.
* Symptomatic central nervous system metastases, carcinomatous meningitis, leptomeningeal disease, or a spinal cord compression that require immediate treatment.
* Clinically significant comorbidities such as significant cardiac or cerebrovascular disease, gastrointestinal disorders that could affect absorption of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Selection Part: Incidence of adverse events | From Date of Randomization up to 16 weeks
  To evaluate the number of participants with adverse events
Dose-Selection Part: Incidence of dose reduction | From Date of Randomization up to 16 weeks
  To evaluate the number of participants reducing the dose of palazestrant
Dose-Selection Part: Incidence of drug discontinuation | From Date of Randomization up to 16 weeks
  To evaluate the number of participants discontinuing palazestrant
Trial: Progression-Free Survival (PFS) | From Date of Randomization until Disease Progression or Death Due to Any Cause (estimated as up to 2 years)
  To compare PFS, based on a Blinded Independent Review Committee (BIRC) assessment, between arms of OP-1250 and standard-of-care treatment. This will be assessed separately in populations of ESR1-mutation detected and ESR1-mutation not detected participants.

SECONDARY OUTCOMES:
Trial: Overall Survival (OS) | From Date of Randomization until Death Due to Any Cause (estimated as up to 4 years)
  To compare OS between arms of OP-1250 and standard-of-care treatment. This will be assessed separately in populations of ESR1 mutation detected and ESR1 mutation not detected participants.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Olema Pharmaceuticals, Inc.
Locations (170):
- United States (38):
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Fountain Valley, California
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Whittier, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Golden, Colorado
  - Clinical Trial Site, Grand Junction, Colorado
  - Clinical Trial Site, Danbury, Connecticut
  - Clinical Trial Site, Newark, Delaware
  - Clinical Trials Site, Jacksonville, Florida
  - Clinical Trial Site, Margate, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Plantation, Florida
  - Clinical Trial Site, Tamarac, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Urbana, Illinois
  - Clinical Trial Site, Baton Rouge, Louisiana
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Saint Louis Park, Minnesota
  - Clinical Trial Site, Lincoln, Nebraska
  - Clinical Trial Site, Farmington, New Mexico
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Port Jefferson Station, New York
  - Clinical Trial Site, Dayton, Ohio
  - Clinical Trial Site, Toledo, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Sayre, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Ogden, Utah
  - Clinical Trial Site, Spokane, Washington
- Argentina (9):
  - Clinical Trial Site, Bahía Blanca, Buenos Aires
  - Clinical Trial Site, Mar del Plata, Buenos Aires
  - Clinical Trial Site, Córdoba, Córdoba Province
  - Clinical Trial Site, San Salvador de Jujuy, Jujuy Province
  - Clinical Trial Site, La Rioja, La Rioja Province
  - Clinical Trial Site, Viedma, Río Negro Province
  - Clinical Trial Site, Rosario, Santa Fe Province
  - Clinical Trial Site, San Miguel de Tucumán, Tucumán Province
  - Clinical Trial Site, Buenos Aires
- Australia (7):
  - Clinical Trial Site, Gosford, New South Wales
  - Clinical Trial Site, Westmead, New South Wales
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Ballarat Central, Victoria
  - Clinical Trial Site, Clayton, Victoria
  - Clinical Trial Site, Shepparton, Victoria
  - Clinical Trial Site, Nedlands, Western Australia
- Belgium (4):
  - Clinical Trial Site, Edegem, Antwerpen
  - Clinical Trial Site, Woluwe-Saint-Lambert, Brussels Capital
  - Clinical Trial Site, Charleroi, Hainaut
  - Clinical Trial Site, Leuven, Vlaams Brabant
- Brazil (7):
  - Clinical Trial Site, Salvador, Estado de Bahia
  - Clinical Trial Site, Belo Horizonte, Minas Gerais
  - Clinical Trial Site, Recife, Pernambuco
  - Clinical Trial Site, Porto Alegre, Rio Grande do Sul
  - Clinical Trial Site, Itajaí, Santa Catarina
  - Clinical Trial Site, Sorocaba, São Paulo
  - Clinical Trial Site, Rio de Janeiro
- Bulgaria (3):
  - Clinical Trial Site, Panagyurishte, Pazardzhik
  - Clinical Trial Site, Sofia, Sofia-Grad
  - Clinical Trial Site, Vratsa, Vratsa
- Canada (4):
  - Clinical Trial Site, Calgary, Alberta
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Czechia (3):
  - Clinical Trial Site, Hradec Králové, Královéhradecký kraj
  - Clinical Trial Site, Nový Jičín, Moravskoslezský kraj
  - Clinical Trial Site, Olomouc, Olomoucký kraj
- France (8):
  - Clinical Trial Site, Bourg-en-Bresse, Ain
  - Clinical Trial Site, Besançon, Doubs
  - Clinical Trial Site, Nantes, Loire-Atlantique
  - Clinical Trial Site, Compiègne, Oise
  - Clinical Trial Site, Clermont-Ferrand, Puy-de-Dôme
  - Clinical Trial Site, Le Mans, Sarthe
  - Clinical Trial Site, Villejuif, Val-de-Marne
  - Clinical Trial Site, Montpellier
- Germany (5):
  - Clinical Trial Site, Karlsruhe, Baden-Wurttemberg
  - Clinical Trial Site, Krefeld, North Rhine-Westphalia
  - Clinical Trial Site, Velbert, North Rhine-Westphalia
  - Clinical Trial Site, Dresden, Saxony
  - Clinical Trial Site, Kiel, Schleswig-Holstein
- Hong Kong (4):
  - Clinical Trial Site, Central, Hong Kong
  - Clinical Trial Site, Kowloon, Hong Kong
  - Clinical Trial Site, Hong Kong
  - Clinical Trials Site, Hong Kong
- Hungary (3):
  - Clinical Trial Site, Pécs, Baranya
  - Clinical Trial Site, Kecskemét, Bács-Kiskun county
  - Clinical Trial Site, Debrecen, Hajdú-Bihar
- Italy (11):
  - Clinical Trial Site, Avellino, Campania
  - Clinical Trial Site, Bologna, Emilia-Romagna
  - Clinical Trial Site, Meldola, Emilia-Romagna
  - Clinical Trial Site, Modena, Emilia-Romagna
  - Clinical Trial Site, Reggio Emilia, Emilia-Romagna
  - Clinical Trial Site, Udine, Friuli Venezia Giulia
  - Clinical Trial Site, Rome, Lazio
  - Clinical Trial Site, Milan, Lombardy
  - Clinical Trial Site, Rozzano, Lombardy
  - Clinical Trial Site, Alessandria, Piedmont
  - Clinical Trial Site, Pavia
- Malaysia (8):
  - Clinical Trials Site, Sungai Petani, Kedah
  - Clinical Trial Site, Kota Bharu, Kelantan
  - Clinical Trial Site, Ipoh, Perak
  - Clinical Trial Site, George Town, Pulau Pinang
  - Clinical Trial Site, Putrajaya, Putramya
  - Clinical Trial Site, Kuching, Sarawak
  - Clinical Trial Site, Petaling Jaya, Selangor
  - Clinical Trial Site, Kuala Lumpur, WP
- Mexico (4):
  - Clinical Trial Site, Zapopan, Jalisco
  - Clinical Trial Site, Monterrey
  - Clinical Trial Site, Oaxaca City
  - Clinical Trial Site, Sinaloa
- Netherlands (2):
  - Clinical Trial Site, Amsterdam, North Holland
  - Clinical Trial Site, Rotterdam, South Holland
- Poland (9):
  - Clinical Trial Site, Skórzewo, Greater Poland Voivodeship
  - Clinical Trial Site, Lublin, Lublin Voivodeship
  - Clinical Trial Site, Lodz, Lódzkie
  - Clinical Trial Site, Otwock, Masovian Voivodeship
  - Clinical Trial Site, Brzozów, Podkarpackie Voivodeship
  - Clinical Trial Site, Rzeszów, Podkarpackie Voivodeship
  - Clinical Trial Site, Gdynia, Pomeranian Voivodeship
  - Clinical Trial Site, Krakow
  - Clinical Trial Site, Wroclaw
- Portugal (4):
  - Clinical Trial Site, Coimbra, Coimbra District
  - Clinical Trial Site, Lisbon, Lisbon District
  - Clinical Trial Site, Matosinhos Municipality, Porto District
  - Clinical Trial Site, Porto, Porto District
- Clinical Trial Site, Mayagüez, Puerto Rico, Puerto Rico
- Romania (7):
  - Clinical Trial Site, Oradea, Bihor County
  - Clinical Trial Site, Brasov, Brașov County
  - Clinical Trial Site, Bucharest, București
  - Clinical Trial Site, Cluj-Napoca, Cluj
  - Clinical Trial Site, Craiova, Dolj
  - Clinical Trial Site, Iași, Iaşi
  - Clinical Trial Site, Timișoara, Timiș County
- South Korea (4):
  - Clinical Trial Site, Suwon, Gyeonggi-do
  - Clinical Trial Site, Busan
  - Clinical Trial Site, Seoul
  - Clinical Trial Site, Suwon
- Spain (11):
  - Clinical Trial Site, Badajoz, Badajoz
  - Clinical Trial Site, Girona, Girona
  - Clinical Trial Site, León, León
  - Clinical Trial Site, Lleida, Lleida
  - Clinical Trial Site, Madrid, Madrid
  - Clinical Trial Site, Pamplona, Navarre
  - Clinical Trial Site, Seville, Sevilla
  - Clinical Trial Site, Valencia, Valencia
  - Clinical Trial Site, Alicante
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Santiago de Compostela
- Taiwan (5):
  - Clinical Trial Site, Changhua
  - Clinical Trial Site, Kaohsiung City
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Tainan
  - Clinical Trial Site, Taipei
- Thailand (4):
  - Clinical Trial Site, Bangkok
  - Clinical Trial Site, Chiang Mai
  - Clinical Trial Site, Samut Sakhon
  - Clinical Trial Site, Songkhla
- United Kingdom (5):
  - Clinical Trial Site, Leicester, Leicestershire
  - Clinical Trial Site, Nottingham, Nottingham
  - Clinical Trial Site, Taunton, Somerset
  - Clinical Trial Site, Bodelwyddan
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pistilli B, Bellet Ezquerra M, Del Mastro L, Sohn J, Schmid P, Meisel J, Chan A, Zheng L, de Kermadec E, McArthur H. OPERA-01: a phase III study of palazestrant for ER+, HER2- advanced breast cancer after CDK4/6 inhibitor therapy. Future Oncol. 2026 Jan;22(2):157-166. doi: 10.1080/14796694.2025.2608863. Epub 2025 Dec 29. PMID 41461598
- See also: Olema Publications — https://olema.com/science/publications